CLINICAL TRIAL: NCT06993883
Title: Use of Venetoclax in AML Patients Retrospective Experience in Sohag Governorate , an Area of Limited Resources in Upper Egypt
Brief Title: Use of Venetoclax , AML , Sohag , Egypt
Acronym: AML
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Walaa Gamal Mohamed Soliman, lecturer of clinical oncology and hemato oncology, Sohag University
Other Study IDs: Soh-Med-25-4-11PD
Record Dates: First submitted 2025-05-13; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: AML (Acute Myelogenous Leukemia)
Keywords: AML; venetoclax; Sohag; Egypt
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- 1st line: newly diagnosed AML patients unfit for aggressive chemotherapy who received reduced intensity protocols plus venetoclax in the 1st line setting.
  Interventions: Drug: Venetoclax
- 2nd line: refractory recurrent AML patients after 1st line chemotherapy who received venetoclax plus 2nd line chemotherapy.
  Interventions: Drug: Venetoclax
- 3rd line: refractory recurrent AML patients after 2 lines chemotherapy who received venetoclax plus 3rd line chemotherapy.
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: Venetoclax — observational study for the result of venetoclax use combined with chemotherapy in AML patients in Sohag governorate

SUMMARY:
retrospective observational study to evaluate the benefit of adding venetoclax to chemotherapy in the first or second line setting in Sohag governorate.

DETAILED DESCRIPTION:
Acute Myeloid Leukaemia (AML) is an aggressive and most common hematologic malignancy in adults with a higher incidence in older adults with a median age of diagnosis of 68 years. It accounts for the largest number of annual deaths from leukaemia. Several new therapies have been approved after many years and are expected to impact patient outcomes, especially in patients aged 60 and above.

The standard treatment strategy for newly diagnosed AML is an intensive curative chemotherapy, and a combination of cytarabine (AraC) and anthracycline is recommended as remission induction therapy. However, many AML patients are ineligible for intensive therapy because of advanced age or co-morbidities. Treatment options are limited for these patients, especially older patients, who account for a large proportion of patients with newly diagnosed AML Venetoclax is an orally available, small-molecule selective B cell leukemia/lymphoma-2 ( BCL-2 ) inhibitor. In two placebo-controlled Phase 3 trials, the safety and efficacy of venetoclax-based therapy were confirmed in treatment-naive patients with AML who were ineligible for intensive chemotherapy owing to advanced age or comorbidities. In the VIALE-A study, the venetoclax plus azacitidine (AZA) arm demonstrated significantly better outcomes compared with the placebo plus AZA arm. In the VIALE-C study, the venetoclax plus LDAC arm did not meet its primary endpoint of a statistically significant improvement in overall survival compared with the placebo plus LDAC arm In November 2018, the US Food and Drug Administration granted accelerated approval for venetoclax in combination with AZA, decitabine or LDAC for the treatment of newly diagnosed AML in adults aged ≥75 years or who have co-morbidities that preclude the use of intensive induction chemotherapy.

Primary refractory disease and relapse remain the main obstacles for cure in AML. In fit patients several options based on higher doses of cytarabine have been published, with complete remission (CR) rates ranging from 40-55%. The BCL2 inhibitor venetoclax has demonstrated impressive antileukemic activity when combined with hypomethylating agents or low-dose cytarabine in newly diagnosed unfit AML patients, the addition of venetoclax to aggressive chemotherapy protocols as a second line in patients with refractory/ relapsed AML patients who are fit for such treatment gives marked advance in treating such difficult situation.

Even in some patients who show great side effects while using first line aggressive treatment , second line use of venetoclax combined with hypomethylating agents as a lower intensity second line option could give a great advance and safe method as a bridge to bone marrow transplantation and cure.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 80 years.
* Pathological confirmation of AML.
* Use of venetoclax plus chemotherapy as a 1st versus 2nd line treatment.

Exclusion Criteria:

age < 18 years age > 80 years other types of acute leukemia

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: observational descriptive study
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
response rate | through the study completion an average 1.5 years

SECONDARY OUTCOMES:
overall survival | 1.5 years
  survival from diagnosis till study end or death

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag Faculty of Medicine, Sohag, Select, Egypt

IPD SHARING:
Plan to Share IPD: Undecided